CLINICAL TRIAL: NCT07354763
Title: Adjustable Temperature Cooler for Cold Static Storage of Donor Hearts for Transplantation
Brief Title: Precise Cooler for Donor Heart Transport
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Dominic Emerson, MD, Associate Surgical Director of Heart Transplant and Mechanical Circulatory Support, Director of Robotic Cardiac Surgery, and Director of the Accreditation Council for Graduate Medical Education Fellowship Program, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00004185
Record Dates: First submitted 2026-01-18; First posted 2026-01-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplantation
Keywords: Donor heart; Heart transplantation; organ procurement; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This study has two study groups. Organ transport using the RYOBI cooler and Organ transport using the Paragonix SherpaPak This means that you will be put in a study group by chance (like flipping a coin). You will be randomly put in one of the above study groups. You will have an equal chance of being placed in any one of the groups described above. A computer will randomly put you in a study group. We do this because no one knows if the results in one study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Organ transport using Standard of Care Paragonix SherpaPak (Active Comparator): In this arm, the organ will be transported using the FDA Approved Sheperpak by Paragonix
  Interventions: Device: Organ transport using SherpaPak
- Organ transport using the RYOBI cooler. (Experimental): In this arm, the organ will be transported using the Ryobi cooler
  Interventions: Device: Ryobi cooler for Organ Transport

INTERVENTIONS:
Device: Organ transport using SherpaPak — Paragonix SherpaPak
  Arms: Organ transport using Standard of Care Paragonix SherpaPak
Device: Ryobi cooler for Organ Transport — This is a temperature-controlled cooler without a gel or ice
  Arms: Organ transport using the RYOBI cooler.

SUMMARY:
The investigators are doing this study to compare approaches to cold storage of donor hearts during transportation. The adjustable temperature RYOBI cooler should allow precise temperature control while reducing environmental waste and providing a cost savings benefit when compared to the commercially available, FDA-approved Paragonix SherpaPak device.

DETAILED DESCRIPTION:
The purpose of this study is to compare outcomes following heart transplant using two different storage devices for transport of the donor heart, an adjustable temperature cooler or a commercially available storage device called the Paragonix SherpaPak.

When a donor heart is identified for transplant, the method of storage during transportation will be randomized to one of two different options for cold storage. All other parts of the participant's care will then continue per usual standard of care. In the thirty days following transplant, the research team will review the participant's medical record to see what medications were used after transplant, what diagnostic studies like echocardiograms showed, and to collect basic information about the participant's medical history.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years old or older are included.
* Individuals undergoing isolated heart transplantation are included.

Exclusion Criteria:

* Any records flagged "break the glass" or "research opt out."
* Any patients undergoing multi-organ transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of primary graft dysfunction | From Randomization to 30 days after heart transplantation
  compare the incidence of primary graft dysfunction between patients randomized to donor heart preservation using the adjustable temperature RYOBI cooler (Model # Pi1824QBT) (n = 40) versus the Paragonix SherpaPak (n = 40) in cases where the anticipated total ischemic time for the graft is between 120 and 240 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No